CLINICAL TRIAL: NCT01285076
Title: Naturalistic Evaluation of Hypoglycemic Events in Diabetic Subjects (NEEDS Study)
Brief Title: Evaluation of Low Blood Sugar Events in Participants With Diabetes (MK-0431-401)
Acronym: NEEDS
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 0431-401
Record Dates: First submitted 2011-01-26; First posted 2011-01-27 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2024-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Enrolled Participants: Adults with Type 2 DM ≥30 years of age who have been treated with SU monotherapy or SU + MF combination therapy for at least 6 months by a cardiologist, nephrologist, neurologist, or family practice doctor.
  Interventions: Other: Other: Retrospective chart review; one participant encounter visit.

INTERVENTIONS:
Other: Other: Retrospective chart review; one participant encounter visit. — Participants will be selected based on medical record review in the office of their treating cardiologist, nephrologist, neurologist, or family practice doctor. Participants will have one encounter visit to fill out questionnaires and have a blood draw and recording of weight, blood pressure and waist circumference.

SUMMARY:
This is a multi-center, observational, retrospective and cross-sectional study to be conducted in a cohort of consecutively selected participants with Type 2 diabetes mellitus (DM) who have been treated with sulphonylurea (SU) monotherapy or SU + metformin (MF) combination therapy by their cardiologist, nephrologist, neurologist, or family practice doctor for at least 6 months prior to Study Enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with Type 2 DM.
* Participants at least 30 years of age at time of Type 2 DM diagnosis.
* Participants treated with SU monotherapy or SU + MF combination therapy for at least 6 months prior to enrollment.
* Participants receiving diabetes care from a cardiologist, nephrologist, neurologist, or family practice doctor for at least 6 months.
* Participants with a clinical record in the health care center.
* Participants in whose medical records a minimum core data set can be found; core data defined as: age, gender, duration of diabetes/age at diagnosis, all glucose-lowering medications (branded and generic names, dosage, dosing frequency, starting and stopping dates) since the start of all antihyperglycemic medications.

Exclusion Criteria:

* Participants with Type 1 DM.
* Participants who are pregnant or with gestational DM.
* Participants receiving any anti-diabetic treatment from an endocrinologist/diabetologist in the previous 6 months.
* Participants requiring daily concomitant usage of insulin.
* Participants receiving any oral diabetes medications other than SU or SU + MF.
* Participants who are already participating in a clinical trial or other clinical study.
* Participants for whom it would be impossible to complete the questionnaire.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with Type 2 DM ≥30 years of age who have been treated with SU monotherapy or SU + MF combination therapy for at least 6 months by a cardiologist, nephrologist, neurologist, or family practice doctor.
Sampling Method: Non-Probability Sample
Enrollment: 834 (Actual)
Dates: Start 2011-01-10 (Actual); Primary Completion 2012-12-27 (Actual); Study Completion 2012-12-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Merck Sharp & Dohme (I.A.) Corp., Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Participants: Adults with Type 2 diabetes mellitus (DM) ≥30 years of age who have been treated with sulphonylurea (SU) monotherapy or SU + metformin (MF) combination therapy for at least 6 months by a cardiologist, nephrologist, neurologist, or family practice doctor.
Period: Overall Study
Arm/Group | All Enrolled Participants
Started | 834
Completed | 834
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 834
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 362
  Male | 472

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Hemoglobin A1C (HbA1C) <7%
Description: HbA1c is measured as a percent.
Time Frame: 6 months
Population: The population analyzed includes only participants with available data.
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 818
participants | 378

2. Primary Outcome: Number of Participants With Hypoglycemic Episodes
Description: Participants self-reported hypoglycemic (low blood sugar) episodes.
Time Frame: 6 months
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 834
participants | 258

3. Secondary Outcome: Score on the Quality of Life (EQ-5D) Questionnaire
Description: The EQ-5D is a standardised instrument for use as a measure of general health outcome. The EQ-5D contains 5 items to be answered using a 3-point Likert scale plus a Visual Analog Scale (VAS). The EQ-5D covers the following dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Total possible score ranges from 0 (worst) to 100 (best).
Time Frame: 1 day (the day of the encounter visit)
Population: The population analyzed includes only participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 823
Score on a scale | 74.2 (14.1)

4. Secondary Outcome: Score on the Treatment Satisfaction Questionnaire for Medication (TSQM)
Description: TSQM is a treatment satisfaction questionnaire. The questionnaire consisted of the following dimensions: side effects (4 items), effectiveness (3 items), convenience (3 items) and global satisfaction scale (3 items). Each dimension was measured as a score on a scale. Total possible score ranges from 0 to 100 with a lower score representing a better quality of life.
Time Frame: 1 day (the day of the encounter visit)
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 834
Score on a scale
  Effectiveness scale | 67.8 (11.7)
  Side effects scale | 75.6 (18.7)
  Convenience scale | 73.5 (12.0)
  Global satisfaction scale | 60.8 (15.4)

5. Secondary Outcome: Number of Adherence Days on the Self-reported Adherence Questionnaire
Description: The self-report adherence questionnaire contains the following items: diabetic diet, exercise, and no missed medication doses during the past week. Total possible score ranges from 0 days (complete non-adherence) to 7 days (complete adherence).
Time Frame: 7 days (during the 7-day period prior to the encounter visit)
Population: All enrolled participants.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 834
Days
  Followed diabetic diet, n=141 | 5.5 (2.3)
  Exercise, n=427 | 5.1 (2.1)
  No missed doses of medication, n=817 | 6.7 (1.1)

6. Secondary Outcome: Experience of Low Blood Sugar (Hypoglycemia) Questionnaire
Description: The experience of low blood sugar questionnaire was developed by the Sponsor to measure the participant's experience of hypoglycemia during the previous 6 months. The questionnaire contains 6 items answered by yes/no or by using a 5-point Likert scale.
Time Frame: 6 months (during the 6-month period prior to the encounter visit)
Population: All enrolled participants.
Measure: Number; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 834
Participants
  With hypoglycemic symptoms | 258 (0.18)
  Mild symptom severity | 155 (0.18)
  Moderate symptom severity | 32 (0.20)
  Severe symptom severity | 47 (0.20)
  Very severe symptom severity | 16 (0.15)
  Unknown symptom severity | 8 (0.11)

7. Secondary Outcome: Score on the Worry Scale of Hypoglycemia Fear Survey (HFS) II
Description: This questionnaire measures a diabetic participant's fear of hypoglycemia. Items were answered using a 5-point Likert scale; range: 1 (never) to 5 (very often). Total possible scores ranged from 18 (least) to 90 (most).
Time Frame: 6 months (during the 6-month period prior to the encounter visit)
Population: The population analyzed includes only participants with available data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 823
Score on a scale | 26.4 (12.2)

8. Secondary Outcome: Experience of Weight Gain Questionnaire
Description: Participants completed a questionnaire regarding weight (wt) gain during the previous year (measured in kilograms[kg]). The questionnaire contained 4 parts: wt gain, subjective severity of wt gain, bothered by wt gain, and difficulty maintaining wt. Percentages presented below are rounded.
Time Frame: 1 year (during the 12-month period prior to the encounter visit)
Population: The population analyzed includes only participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 202
Percentage of participants
  Wt gain <5 kg | 89.6
  Wt gain 5-9 kg | 6.4
  Wt gain 10-15 kg | 1.5
  Wt gain >15 kg | 2.5
  Subjective severity of wt gain: very mild, n=122 | 36.1
  Subjective severity of wt gain: mild, n=122 | 32.0
  Subjective severity of wt gain: moderate, n=122 | 19.7
  Subjective severity of wt gain: severe, n=122 | 9.0
  Subjective severity of wt gain: very severe, n=122 | 3.3
  Bothered by wt gain: not at all, n=122 | 36.1
  Bothered by wt gain: a little bit, n=122 | 27.0
  Bothered by wt gain: somewhat, n=122 | 26.2
  Bothered by wt gain: very, n=122 | 8.2
  Bothered by wt gain: extremely, n=122 | 2.5
  Difficulty maintaining wt: not at all, n=122 | 29.5
  Difficulty maintaining wt: a little bit, n=122 | 25.4
  Difficulty maintaining wt: somewhat, n=122 | 30.3
  Difficulty maintaining wt: very, n=122 | 13.1
  Difficulty maintaining wt: extremely, n=122 | 1.7

9. Secondary Outcome: Fear of Weight Gain Questionnaire
Description: Participants completed a questionnaire regarding their fear of wt gain during the previous year. The questionnaire contained 3 parts: worried about wt gain, worried that diabetic treatment causes wt gain (worried diab tx and wt gain), and worried about not being able to stabilize wt (worried not stabilize wt).
Time Frame: 1 year (during the 12-month period prior to the encounter visit)
Population: The population analyzed only includes participants with available data.
Measure: Number; unit: Percentage of participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 803
Percentage of participants
  Worried about wt gain: never | 49.2
  Worried about wt gain: rarely | 21.3
  Worried about wt gain: sometimes | 15.7
  Worried about wt gain: often | 8.2
  Worried about wt gain: almost always | 5.6
  Worried diab tx and wt gain: never; n=799 | 61.2
  Worried diab tx and wt gain: rarely; n=799 | 20.2
  Worried diab tx and wt gain: sometimes; n=799 | 11.6
  Worried diabetic tx and wt gain: often; n=799 | 4.4
  Worried diab tx and wt gain: almost always; n=799 | 2.6
  Worried not stabilize wt: never; n=799 | 54.8
  Worried not stabilize wt: rarely; n=799 | 20.9
  Worried not stabilize wt: sometimes; n=799 | 13.3
  Worried not stabilize wt: often; n=799 | 7.5
  Worried not stabilize wt: almost always; n=799 | 3.5

10. Secondary Outcome: Self-reported Barrier Questionnaire
Description: The self-report barrier questionnaire contains 4 items: difficulty filling prescriptions, unsure about physician instructions, unable to follow plan for diabetes, and bothered by adverse effects during the prior month.
Time Frame: 30 days (during the 30-day period prior to the encounter visit)
Population: All enrolled participants.
Measure: Number; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 834
Participants
  Any of the barriers listed below | 520
  Barrier: difficulty filling prescriptions | 174
  Barrier: unsure about physician instructions | 393
  Barrier: unable to follow plan for diabetes | 436
  Barrier: bothered by adverse effects | 137

ADVERSE EVENTS:
Time Frame: Up to 24 hours following the encounter visit
Arm/Group | All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 0/834
Other Adverse Events (participants affected / at risk) | 0/834

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator can publish the study results only following the sponsor's review and approval.